CLINICAL TRIAL: NCT02822768
Title: Is Routine Packing of Cutaneous Abscesses Necessary?
Brief Title: Packing Versus no Packing for Cutaneous Abscess
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016052
Record Dates: First submitted 2016-06-30; First posted 2016-07-04 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Cutaneous Abscess
MeSH Terms: interventions — Drug Packaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Packing (Active Comparator): The patient is to have a long piece of gauze within the abscess cavity in an attempt to keep it open and allow purulent material to continue to drain after the initial incision and release of purulent material has been performed.
  Interventions: Procedure: Packing
- No packing (Placebo Comparator): The patient is not to have packing of the abscess as part of the incision and drainage procedure
  Interventions: Other: No packing

INTERVENTIONS:
Procedure: Packing — The patient will receive packing as part of their wound care
  Arms: Packing
Other: No packing — The patient will not receive packing as part of their wound care
  Arms: No packing

SUMMARY:
The goal of this study is to examine patients undergoing incision and drainage of cutaneous abscesses to determine if routine packing of the abscess cavity affects the need for further interventions such as repeat incision and drainage, antibiotic administration or hospital admission.

DETAILED DESCRIPTION:
Study protocol:

1. Identification of a patient with a cutaneous abscess requiring incision and drainage
2. Written consent obtained from the patient
3. Study materials will be obtained

   * Enrolling physician fills out pre-procedure information (see data sheet)
   * Enrollment data sheet has instructions indicating whether patient is to receive packing or not

     * Use of random number generator to randomize all packets
   * Provider does abscess incision and drainage with or without packing according to the instructions
   * Enrolling physician fills out post-procedure information (see data sheet)
   * Patient returns within 48 hours for wound check with removal of packing if performed
   * Research coordinator or study physician calls the patient within 14 and 30 days after the procedure for follow-up

     * Information from a return visit and/or the telephone follow-up

ELIGIBILITY:
Inclusion Criteria:

1. All patients 18 years of age and above
2. Patients that require a cutaneous abscess incision and drainage
3. English-speaking subjects only

Exclusion Criteria:

1. Unable to return for 48-hour follow-up.
2. Patients being admitted to the hospital or going to the operating room for incision and drainage
3. Pregnant patients
4. Patients less than 18 years of age
5. Prisoners or persons in police custody
6. Patients with infected bursa
7. Non-English speaking subjects

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2016-08 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients needing further treatment | 14 days
  follow-up call to determine if patient required further treatment beyond routine care

SECONDARY OUTCOMES:
Visual Analog Scale for Pain (VAS pain) post procedure | 14 days
  Measure pain score after procedure

CONTACTS AND LOCATIONS:
Overall Officials: Michael Darracq, MD, MPH, Principal Investigator — UCSF - Fresno
Locations (1):
- Community Regional Medical Center, Fresno, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Malley GF, Dominici P, Giraldo P, Aguilera E, Verma M, Lares C, Burger P, Williams E. Routine packing of simple cutaneous abscesses is painful and probably unnecessary. Acad Emerg Med. 2009 May;16(5):470-3. doi: 10.1111/j.1553-2712.2009.00409.x. Epub 2009 Apr 10. PMID 19388915
- [Background] Abraham N, Doudle M, Carson P. Open versus closed surgical treatment of abscesses: a controlled clinical trial. Aust N Z J Surg. 1997 Apr;67(4):173-6. doi: 10.1111/j.1445-2197.1997.tb01934.x. PMID 9137156
- [Background] Stewart MP, Laing MR, Krukowski ZH. Treatment of acute abscesses by incision, curettage and primary suture without antibiotics: a controlled clinical trial. Br J Surg. 1985 Jan;72(1):66-7. doi: 10.1002/bjs.1800720125. PMID 3881155
- [Background] Barnes SM, Milsom PL. Abscesses: an open and shut case! Arch Emerg Med. 1988 Dec;5(4):200-5. doi: 10.1136/emj.5.4.200. PMID 3069102
- [Background] Simms MH, Curran F, Johnson RA, Oates J, Givel JC, Chabloz R, ALexander-Williams J. Treatment of acute abscesses in the casualty department. Br Med J (Clin Res Ed). 1982 Jun 19;284(6332):1827-9. doi: 10.1136/bmj.284.6332.1827. PMID 6805714
- [Background] Sorensen C, Hjortrup A, Moesgaard F, Lykkegaard-Nielsen M. Linear incision and curettage vs. deroofing and drainage in subcutaneous abscess. A randomized clinical trial. Acta Chir Scand. 1987 Nov-Dec;153(11-12):659-60. PMID 3324596
- [Background] Tonkin DM, Murphy E, Brooke-Smith M, Hollington P, Rieger N, Hockley S, Richardson N, Wattchow DA. Perianal abscess: a pilot study comparing packing with nonpacking of the abscess cavity. Dis Colon Rectum. 2004 Sep;47(9):1510-4. doi: 10.1007/s10350-004-0620-1. Epub 2004 Jul 8. PMID 15486749